CLINICAL TRIAL: NCT00001233
Title: A Longitudinal Study of Children at Risk for Disruptive Behavior Disorders: Transitions From Early Childhood to Middle Childhood and Adolescence
Brief Title: Study of Children at Risk for Disruptive Behavior Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 880217; 88-M-0217
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders; Child Behavior Disorders; Passive-Aggressive Personality Disorder
Keywords: Adolescence; Aggressivity; Anger; Developmental Psychopathology; Disruptive Behavior Disorders; Early Onset Aggression; Emotion Regulation; Family Violence; Preschool Conduct Problems
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Child Behavior Disorders; Passive-Aggressive Personality Disorder; Emotional Regulation

SUMMARY:
A conduct disorder is characterized by repetitive and persistent patterns of behavior where the basic rights of others and rules are violated.

This study investigates characteristics of children and their surroundings (environments) that place them at risk for the development of disruptive behavior disorders and associated disorders of anxiety and mood. Children ages 4 - 5 with moderate (subclinical) and severe (clinical) rates of misconduct during the preschool period are compared to low risk children. Children and their families were recruited from 1989-1991 and are being studied at five specific times:

1. Preschool (4 - 5 years)
2. Early childhood (6 - 7 years)
3. Middle childhood (9 - 10 years)
4. Early adolescence (13 - 14 years)
5. Mid-adolescence (15 - 16 years)

Researchers will look closely at biological, intellectual, emotional, and behavioral factors that are thought to protect against and/or increase the risk of developing a conduct problem. These factors have been studied in older children and are shown to be associated with disruptive behavior disorders.

The goals of this research study are;

1. Create a database showing the characteristics of the development of disruptive behavior problems.
2. Identify the key risk and protective factors that contribute to the stability or change in behavior problems over time.
3. Identify the ways that children interact socially and relate them to the possibility of developing a problem of behavior.
4. Identify how experiences and the emotions associated with experiences may play a role in the development of related psychiatric conditions, like depression and anxiety.
5. Establish measures of the different components of negative emotions associated with disruptive/antisocial, anxiety, and mood disorders.

DETAILED DESCRIPTION:
This study investigates characteristics of children and their environments that place them at risk for the development of disruptive behavior disorders and co-morbid internalizing problems (anxiety and mood disorders). Children ages 4-5 with moderate (subclinical) and high (clinical) rates of misconduct during the preschool period are compared with low risk children. Children and their families are studied again at four later time points: (a) early childhood (6-7 yrs.), (b) middle childhood (9-10 yrs.), (c) early adolescence (13-14 yrs.), and (d) mid-adolescence (15-16 yrs.). Assessments of children include dimensions of biological, cognitive, affective, emotional and behavioral functioning, that have been identified in research with older children as putative risk and protective factors in the development of conduct problems. Socialization experiences within and outside the family, also hypothesized to influence developmental trajectories are examined. Currently, Time 4 assessments are being conducted, with three-quarters of the research subjects tested. Behavior problems show significant stability across the first three time periods. However, some children improve over time, changes that result, in part, from more optimal environmental conditions. Different patterns of emotion dysregulation, ANS, and HPA activity in antisocial preschool children predict different types of externalizing problems at later time points. Behavior problems and their correlates differ for young disruptive boys and girls: Oppositional, aggressive girls are more likely to have co-morbid internalizing problems, and emotion regulation patterns that may decrease risk for continued antisocial behavior, but increase risk for depression and anxiety later in development.

ELIGIBILITY:
Preschool age children with conduct problems and normal preschool age children used for control.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 1988-12; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Achenbach TM, Edelbrock CS. Behavioral problems and competencies reported by parents of normal and disturbed children aged four through sixteen. Monogr Soc Res Child Dev. 1981;46(1):1-82. PMID 7242540
- [Background] Achenbach TM, Edelbrock CS. The classification of child psychopathology: a review and analysis of empirical efforts. Psychol Bull. 1978 Nov;85(6):1275-1301. No abstract available. PMID 366649
- [Background] Cole PM, Zahn-Waxler C, Fox NA, Usher BA, Welsh JD. Individual differences in emotion regulation and behavior problems in preschool children. J Abnorm Psychol. 1996 Nov;105(4):518-29. PMID 8952185